CLINICAL TRIAL: NCT06160336
Title: Use of Transcutaneous Electrical Stimulation for Restoring Somatotopic Sensory Feedback in Lower Limb Amputees
Brief Title: Transcutaneous Electrical Stimulation in Lower Limb Amputees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Campus Bio-Medico University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SENSE
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Lower Limb Amputation
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TENS group (Experimental)
  Interventions: Other: Transcutaneous Electrical Nerve Stimulation

INTERVENTIONS:
Other: Transcutaneous Electrical Nerve Stimulation — Phase 1: Participants undergo a comprehensive assessment in a single experimental session (mapping session) aimed at mapping the regions and sensations that can be electrically stimulated. This mapping protocol is conducted on both the intact and amputated limbs.
  Phase 2: This phase comprises a 4-week experimental protocol, including:
  1. four mapping sessions conducted at the onset of each week, where the protocol is randomly applied to the participant's intact and amputated limb.
  2. three stimulation sessions held over three consecutive days in the initial week to assess the participant's ability to discern stimuli of varying intensities.
  3. ten sessions utilizing an end-effector gait rehabilitation robot, aiming to train the participant in walking using the proposed sensory feedback restoration system based on TENS under controlled and repeatable experimental conditions.

SUMMARY:
Current lower limb prostheses support ambulation by absorbing and stabilizing positions during walking. Users of lower limb prostheses rely solely on sensory information provided by the contact between the socket and the residual limb. Restoring sensory feedback could potentially improve their quality of life and participation in daily activities. Despite a high incidence of lower limb amputations, there are few studies in the literature addressing the restoration of sensory feedback in lower limb amputees, particularly studies utilizing invasive techniques. In an effort to overcome these limitations, various non-invasive methods have been tested. Despite resulting benefits such as improved gait symmetry and stability, most non-invasive stimulation systems are non-somatotopic, failing to generate a sensation referred to the patient's missing limb. From the literature, Transcutaneous Electrical Nerve Stimulation (TENS) emerges as a very promising non-invasive and somatotopically-based sensory feedback approach, capable of inducing sensations referred to the amputees' phantom limb.

Therefore, the proposed study will involve the use of TENS as a means to stimulate sensitivity and prevent perceptual disturbances associated with the interruption of peripheral nerve structures occurring in individuals undergoing amputation. These disturbances, besides influencing the development of symptoms characterized by neuropathic pain, can impact prosthesis management.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 80 years;
2. unilateral transtibial amputation or transfemoral amputation at least two months prior the study;
3. stable clinical conditions;
4. skin integrity;
5. absence of cognitive deficits.

Exclusion Criteria:

1. bilateral amputation;
2. open wounds or sores on the residual limb;
3. cognitive deficits;
4. pregnancy;
5. presence of implanted medical device (e.g., cardiac defibrillators, pacemakers or infusion pumps);
6. refusal to sign the informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-03-14 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2023-08-04 (Actual)

PRIMARY OUTCOMES:
Electrical Sensation Mapping Questionnaire | Baseline
  It is an ad-hoc questionnaire designed for comprehensive characterization of sensations elicited through TENS. This includes perceptual thresholds, referred sensations (evaluated for naturalness, depth, pain, intensity, and quality), sensitivity, size, and similarity of the activated areas.
  The questionnaire incorporates: a five-point scale assessing naturalness from unnatural to natural, a metric to determine the sensation's location (i.e., superficial and/or deep), a scale from 0 to 10 measuring the intensity and pain levels of the sensation, and multiple choice options to describe the quality (touch/pressure, pinch, vibration, tugging, tingling, burning, hot, cold, ankle flexion, ankle extension, toe flexion, toe extension, and none)

SECONDARY OUTCOMES:
Changes in body weight distribution between legs during gait | Baseline; after a 1-month intervention
  Assessment of the force exerted on the ground during walking using an ad-hoc developed insole equipped with sensors, designed to be inserted under the participant's prosthetic foot.
Changes in gait symmetry | Baseline; after a 1-month intervention
  Evaluation of the symmetry between the intact and the amputated limbs based on spatio-temporal gait parameter, measured using an optoelectronic system
Changes in Pain Intensity (NRS) | Baseline; after a 1-month intervention
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale, from 0 (no pain) to 10 (worst pain imaginable)
Changes in Neuropathic Pain (NPSI) | Baseline; after a 1-month intervention
  The NPSI is one of the most extensively used instruments for assessing the intensity of neuropathic pain symptoms. It consists of 10 items corresponding to sensory descriptors that can be grouped into 5 dimensions: spontaneous burning pain (burning), spontaneous pressing pain (pressing), paroxysmal pain (paroxysmal), evoked pain (evoked), and paresthesia/dysesthesia.
  Each dimension can be scored between 0 and 10. In addition, a final score, equivalent to the total of the 10 descriptors and ranging from 0 (best) to 100 (worst), can be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Don Carlo Gnocchi, Centro Santa Maria della Provvidenza, Roma, Italy